CLINICAL TRIAL: NCT00057278
Title: Gabapentin in Fibromyalgia Trial (GIFT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR22264; NIAMS-089
Record Dates: First submitted 2003-03-28; First posted 2003-03-31 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Fibromyalgia
Keywords: Gabapentin
MeSH Terms: conditions — Fibromyalgia | interventions — Gabapentin

INTERVENTIONS:
Drug: gabapentin

SUMMARY:
This study will assess the safety and effectiveness of the drug gabapentin in reducing pain associated with primary fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia, a chronic musculoskeletal pain disorder of unknown etiology, is characterized by widespread musculoskeletal pain, fatigue, and multiple tender points; the disease affects 3 to 6 million Americans. A person is considered to have fibromyalgia if he or she has widespread pain in combination with tenderness in at least 11 of 18 specific tender point sites.

Treatment of fibromyalgia requires a comprehensive approach and includes aerobic exercise, heat and massage, antidepressant medications, and relaxation. Gabapentin, a medication used to treat seizures, has been shown to work on pain transmission pathways and may relieve the pain associated with fibromyalgia. This study will assess the efficacy of gabapentin in reducing pain severity in fibromyalgia as measured by the average pain item of the Brief Pain Inventory (BPI) score.

Patients will be randomized to receive gabapentin or placebo. The gabapentin dose will be titrated for persisting symptoms and as tolerated during the first 6 weeks of the study, reaching final doses between 1800 mg/day and 2400 mg/day. Patients will then continue on the final dose for the remaining 6 weeks of the study. Following completion of the 12 week treatment phase, patients will be tapered off of the medication over 1 week.

The effectiveness of gabapentin will be assessed using the BPI. The BPI is a self-administered questionnaire that measures the severity of pain and the interference of pain on function over the past 24 hours. Other assessments will include the total Fibromyalgia Impact Questionnaire (FIQ) score; six 11-point Likert-type scales in the FIQ that measure pain, fatigue, morning tiredness, stiffness, anxiety, and depression; the mean tender point pain threshold; Clinical Global Impression of Severity (CGI-Severity); Patient Global Impression of Improvement (PGI-Improvement); the Short-form McGill Pain Questionnaire (SF-MPQ); the Medical Outcomes Study Short Form-36 (SF-36); the Montgomery Asberg Depression Rating Scale (MADRS); and the Medical Outcomes Sleep Scale (MOS-Sleep).

ELIGIBILITY:
Inclusion Criteria:

* Primary fibromyalgia as defined by the American College of Rheumatology (ACR)
* Score greater than 4 on the average pain item of the BPI at screening
* Ability to understand and cooperate with study procedures
* Acceptable methods of contraception

Exclusion Criteria:

* Unwillingness or inability to provide written informed consent.
* Lifetime history of psychosis, hypomania or mania, epilepsy, or dementia
* History of seizures or status epilepticus
* DSM-IV diagnosis of alcohol or substance dependence with the exception of nicotine dependence within 6 months prior to screening visit
* A positive urine drug screen for any substances of abuse or excluded medication. (NOTE: If the participant has a positive drug screen at Visit 1 for an excluded medication that may not have had an adequate wash-out period, a retest may be performed prior to Visit 2. If the retest is positive, the participant will be excluded.)
* Serious suicide risk
* Treatment refractory in the opinion of study official
* Pregnant or breastfeeding
* Clinically unstable medical or psychiatric condition that could interfere with the absorption, metabolism, excretion, or safety of gabapentin or interfere with the assessment of disease severity
* Thyroid-stimulating hormone (TSH) concentrations outside the range of 0.30-8.0 UlU/mL. (NOTE: Participants who have been on a stable dose of thyroid supplementation for at least the past 3 months, have medically appropriate TSH values, and are clinically euthyroid may participate in the study.)
* Any screening laboratory assay that is outside of the local laboratories' normal range by more than 20% or is deemed to be a clinically significant abnormality by the investigator, with the exception of liver function tests (AST, ALT, alkaline phosphatase) which must be within 1.5 X upper limit of normal
* Inability to exclude traumatic injury, regional or structural rheumatic disease, or infectious arthropathy as the etiology of their relevant symptoms and that would interfere with interpretation of outcome measures (e.g., osteoarthritis, bursitis, tendonitis)
* History of an autoimmune disease or inflammatory arthritis, such as systemic lupus erythematosis (SLE) or rheumatoid arthritis (RA).
* An abnormal Westergren erythrocyte sedimentation rate (e.g., ESR > 40 mm/min)
* An abnormal antinuclear antibody (ANA > 1:160) or rheumatoid factor (RF >15 IU/ml)
* Treatment with a monoamine oxidase inhibitor, tricyclic, SSRI antidepressant (with the exception of fluoxetine), or lithium within 2 weeks prior to beginning study medication
* Treatment with fluoxetine within 30 days prior to beginning study medication
* Treatment with analgesic medication (with the exception of acetaminophen and over-the-counter NSAIDs) within 1 week prior to beginning study medication
* Treatment with any other excluded medications that cannot be discontinued at the screening visit (see Table 2 for a list of excluded medications)
* Previous treatment with gabapentin
* Previous treatment with pregabalin
* Treatment with any other investigational medications within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) average pain item

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire
Mean Tender Point Pain Threshold
McGill Pain Questionnaire
Clinical Global Impression of Severity
Patient Global Impression of Improvement
Montgomery-Asberg Depression Rating Scale (MADRS)
Medical Outcomes Study Short Form-36 (SF-36)
Medical Outcomes Sleep Scale (MOS-Sleep)
Fibromyalgia Rating Scale (FRS)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley M. Arnold, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - McLean Hospital/Harvard Medical School (must live in the Boston, MA area), Belmont, Massachusetts
  - Newton-Wellesley Hospital (must live in the Boston, MA area), Newton, Massachusetts
  - University of Cincinnati College of Medicine, Department of Psychiatry (must live in the Cincinnati, OH area), Cincinnati, Ohio